CLINICAL TRIAL: NCT06104930
Title: Plasma Extracellular Vesicles in Meningioma Patients Following Radiotherapy as Liquid Biopsy
Brief Title: Plasma Extracellular Vesicles in Meningioma Patients
Acronym: MOLI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Department head, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RADONK-MOLI-2023
Record Dates: First submitted 2023-10-11; First posted 2023-10-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Intervention Model Description: Prospective Explorative Biomarker Study / Investigator-Initiated Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Explorative biomarker study — Analysis of blood biomarker

SUMMARY:
While surgical resection remains the primary treatment approach for symptomatic or growing meningiomas, radiotherapy represents an auspicious alternative in patients with meningiomas not safely amenable to surgery. Biopsies are often omitted in light of potential postoperative neurological deficits, resulting in a lack of histological grading and (molecular) risk stratification. In this prospective explorative biomarker study, extracellular vesicles in the bloodstream will be investigated in patients with macroscopic meningiomas to identify a biomarker for molecular risk stratification and disease monitoring.

DETAILED DESCRIPTION:
In total, 60 patients with meningiomas and an indication of radiotherapy (RT) and macroscopic tumor on the planning MRI will be enrolled. Blood samples will be obtained before the start, during, and after radiotherapy, as well as during clinical follow-up every 6 months. Extracellular vesicles will be isolated from the blood samples, quantified and correlated with the clinical treatment response or progression. Further, nanopore sequencing-based DNA methylation profiles of plasma EV-DNA will be generated for methylation-based meningioma classification.

This study will explore the dynamic of plasma EVs in meningioma patients under/after radiotherapy, with the objective of identifying potential biomarkers of (early) tumor progression. DNA methylation profiling of plasma EVs in meningioma patients may enable molecular risk stratification, facilitating a molecularly-guided clinical management in meningioma patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* confirmed meningioma (histologically or MRI/DOTATOC-PET CT)
* macroscopic tumor in MRI (either as definitive RT, or following subtotal resection or relapse)
* indication for radiotherapy
* completed wound healing after surgical intervention)
* Alter ≥ 18 Jahre
* Karnofsky Performance Score ≥ 60%
* written informed consent
* ability of subject to understand character and individual consequences of the trial
* adequate contraception for women of childbearing potential

Exclusion Criteria:

* previous or known tumor diseases < 5 years ago
* previous (cerebral) radiotherapy
* simultaneous chemo/immunotherapy
* evidence that the patient cannot adhere to the study protocol (e.g., non-compliance)
* the refusal of patients to participate in the study
* participation in another clinical study or observation period in a competing trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
dynamic of plasma EVs | until 2 years follwoing radiotherapy
  Change of amount of plasma EVs in meningioma patients compared to sample taken before radiotherapy

SECONDARY OUTCOMES:
progession-fee survival | until 2 years follwoing radiotherapy
  number of patients without tumor progress
overall survival | until 2 years follwoing radiotherapy
  number of alive patients

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Heidelberg, Radiation Oncology, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No